CLINICAL TRIAL: NCT05364099
Title: Suprascapular Nerve Block for Treatment of Shoulder Pain in Individuals With Spinal Cord Injuries
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to feasibly complete study.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Timothy Tiu, Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220014
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Chronic Shoulder Pain
Keywords: Overuse Shoulder Syndrome
MeSH Terms: interventions — Lidocaine; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Suprascapular Nerve Block in Participants with Spinal Cord Injuries (SCI) Group (Experimental): Participants in this group will receive standard of care (SOC) suprascapular nerve block using a mixture of Lidocaine and Triamcinolone.
  Interventions: Drug: Lidocaine 1% Injectable Solution; Drug: Triamcinolone Injection; Procedure: Suprascapular Nerve Block

INTERVENTIONS:
Drug: Lidocaine 1% Injectable Solution — 2.5 ml of 1% Lidocaine will be administered via injection in suprascapular nerve in the suprascapular notch
Drug: Triamcinolone Injection — 0.5 ml 40mg/ml Triamcinolone will be administered via injection in suprascapular nerve in the suprascapular notch
Procedure: Suprascapular Nerve Block — This procedure involves injection of a lidocaine and triamcinolone mixture into the suprascapular nerve in the suprascapular notch using ultrasound guidance for proper placement of drugs.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of using suprascapular nerve block for individuals with chronic spinal cord injury who have chronic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-70 years of age, inclusive. 2 Neurological impairment secondary to SCI that occurred at least twelve (12) months prior to the Screening Visit; neurological level of injury between C6 and L5, inclusive.

3. Non-ambulatory, except for exercise or therapy purposes. 4. Uses a manual wheelchair. 5 History of chronic shoulder pain for ≥6 months that has been unresponsive to conservative treatment (e.g. physical therapy, pharmacological agents), and is rated as ≥4 out of 10 on an 11-point Numeric Rating Scale (NRS) (0 = "no pain"; 10 = "most intense pain imaginable") for average shoulder pain intensity during the week leading up to the Screening Visit.

6. Able and willing to comply with the protocol. 7. Able to give voluntary informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

1. Contra-indications to the procedure (e.g. infection, coagulopathy)
2. History of active cancer within 5 years
3. Adhesive capsulitis
4. Prior history of regenerative medicine intervention
5. Glucocorticoid injection within the past four weeks
6. Any medical condition, including psychiatric illness, which would interfere with the interpretation of the study results or the conduct of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants at each Global Satisfaction Rating (GSR) | 1 month post procedure
  Global Satisfaction Score is rated as: Very Dissatisfied, Dissatisfied, Neutral, Satisfied and Very Satisfied
Number of participants reporting treatment related adverse events | Up to 12 months
  As per treating physician evaluation of participant adverse events related to the intervention

SECONDARY OUTCOMES:
Number of participants at each Global Satisfaction Rating | Up to 12 months post procedure
  Global Satisfaction Score is rated as: Very Dissatisfied, Dissatisfied, Neutral, Satisfied and Very Satisfied
Change in NRS scores | Baseline, 12 months
  Numerical rating scores (NRS) ranges from 0 to 10 with highest score indicating the maximum pain and the lowest score indicating the lowest amount of pain.
Change in DASH Questionnaire scores | Baseline, 12 months
  Disability of the Arm, Shoulder, and Hand (DASH) questionnaire is a 30-item questionnaire evaluating the ability of the patient to perform upper extremity activities. The questions are measured on a 5-point Likert scale with 1 being no difficulty and 5 bring unable to perform the activity.
Change in BPI-I scores | Baseline, 12 months
  Brief Pain Inventory pain Interference items (BPI-I) scores ranges from 0-10 with the higher scores indicating greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Tiu, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No